Protocol Number: VX17-445-102

#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Statistical Analysis Plan (Methods)

Protocol Number VX17-445-102 Version 3.0 (Final and Interim Analysis)

A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the *F508del* Mutation and a Minimal Function Mutation (F/MF)

**Authors of SAP:** 

Version: 1.0
Version Date of SAP: 25 September 2018

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, Massachusetts 02210-1862


This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# 2 TABLE OF CONTENTS

| I | Title Page | | |
|---|---|---|---|
| 2 | Table of Contents | | |
| 3 | Mo | difications | . : |
| | 3.1 | Modifications to the Approved Clinical Study Protocol | |
| | 3.2 | Modifications to the Approved Statistical Analysis Plan | |
| | 3.3 | Modifications to the Approved DMC Charter | |
| 4 | | roduction | |
| 5 | | dy Objectives | |
| | 5.1 | Primary Objective | |
| | 5.2 | Secondary Objectives | |
| 6 | | dy Endpoints | |
| | 6.1 | Efficacy and Pharmacodynamic Endpoints | |
| | 6.1 | | |
| | 6.1 | | |
| | 6.2 | Safety Endpoints | |
| | 6.3 | Pharmacokinetic Endpoint. | • |
| 7 | Stu | dy Dosign | |
| / | 7.1 | dy Design Overall Design | |
| | 7.1 | Sample Size and Power | |
| | 7.3 | Randomization. | |
| | 7.4 | Blinding and Unblinding | |
| | 7.5 | Interim Analysis | |
| 8 | | alvsis Sets. | |
| • | 8.1 | All Subjects Set | |
| | 8.2 | Full Analysis Set. | |
| | 8.3 | Safety Set | |
| | 8.4 | Analysis Sets for IA. | |
| | 8.4 | | |
| | 8.4 | · | |
| 9 | Sta | tistical Analysis | |
| | 9.1 | General Considerations | 1 |
| | 9.2 | Background Characteristics | 12 |
| | 9.2 | .1 Subject Disposition | 12 |
| | 9.2 | .2 Demographics and Baseline Characteristics | 13 |
| | 9.2 | | |
| | 9.2 | .4 Prior and Concomitant Medications | 14 |
| | 9.2 | .5 Study Drug Exposure | 14 |
| | 9.2 | .6 Study Drug Compliance | 15 |
| | 9.2 | 1 | |
| | 9.3 | Efficacy Analysis | |
| | 9.3 | | |
| | | 9.3.1.1 Definition of Variables | |
| | ( | 9.3.1.2 Primary Analysis | 16 |

| 9.3.1.3 Supportive Analyses | |
|---|---|
| 9.3.1.4 Sensitivity Analyses | |
| 9.3.1.5 Subgroup Analysis | |
| 9.3.2 Analysis of Key Secondary Variable | s |
| · | |
| ± • • | les20 |
| • | iables |
| 9.3.4.3 Analysis of Additional Variables | s for Pulmonary Exacerbations and |
| taran da antara da a | |
| <u> </u> | $\sim$ 26 |
| $oldsymbol{arepsilon}$ | $\sim$ 26 |
| <u> </u> | |
| • | |
| * * * | est |
| <del>_</del> | |
| 10 SUMMARY OF INTERIM AND DMC AN | ALYSIS |
| 10.1 Interim Analysis | |
| • | |
| | 28 |
| 10.1.2.2 Demographics and Baseline Cha | racteristics |
| | riable29 |
| | cacy Variable |
| · | |
| 10.2 DMC Analysis | |
| 10.2.1 DMC Safety/Efficacy Review | |
| 12 List of Appendices | |
| Annendix A: Analysis Visit Windows for Safet | |

| Appendix B: Imputation Rules for Missing Prior/Concomitant Medication Dates | 37 |
|---|---|
| Appendix C: Details of GLI Equations for Calculating ppFEV <sub>1</sub> | |
| Appendix D: Steps for Multiple Imputation | |
| Appendix E: Imputation Rules for Missing AE dates | |
| Appendix F: Criteria for Threshold Analysis | |
| Appendix G: Adverse Events of Special Interest | |

# 3 MODIFICATIONS

- **3.1** Modifications to the Approved Clinical Study Protocol Not Applicable.
- 3.2 Modifications to the Approved Statistical Analysis Plan

This is the 1<sup>st</sup> version of Statistical Analysis Plan for the final and interim analysis.

**3.3 Modifications to the Approved DMC Charter** Not Applicable.

#### 4 INTRODUCTION

This statistical analysis plan (SAP) for the interim and final analysis is based on the most recent approved clinical study protocol (CSP), electronic case report form (eCRF), and eCRF completion guidelines.

This SAP (Methods) documents the planned statistical analyses of efficacy endpoints and safety endpoints for the interim analysis (IA) and the final analysis. It also documents analyses for additional efficacy and safety variables not specified in the protocol, which will provide supportive information for the scientific understanding of the study drug entity.

The pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of VX-445 in the population heterozygous for the *F508del* mutation and a minimal function mutation will also be evaluated in the study. Selected analyses related to sweat chloride will be documented in this SAP, other PK and PD analyses will be documented separately in the clinical pharmacology analysis plan (CPAP) for the study.

This SAP (Methods) will be finalized and approved prior to IA data lock and treatment unblinding for the IA. Any revisions to the approved SAP will be documented and approved in an amendment to the SAP.

The Vertex Biometrics Department will perform the statistical analysis for the final analysis and prepare the analysis package for the IA; SAS (Version 9.4 or higher) will be used to generate all statistical outputs (tables, figures, listings, and datasets).

appointed as the independent biostatistician, will perform the IA according to the DMC SAP and present the results to the DMC. If the DMC declares that the study has crossed the efficacy boundary, a limited Vertex unblinded team (independent of the study team) may be unblinded to the study and prepare for regulatory submission(s) based on the IA.

#### 5 STUDY OBJECTIVES

#### 5.1 Primary Objective

To evaluate the efficacy of VX-445 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are heterozygous for *F508del* and a minimal function mutation (F/MF subjects)

# 5.2 Secondary Objectives

- To evaluate the safety of VX-445 in TC with TEZ and IVA
- To evaluate the pharmacodynamics (PD) of VX-445 in TC with TEZ and IVA
- To evaluate the pharmacokinetics (PK) of VX-445, TEZ, and IVA when administered in TC

#### 6 STUDY ENDPOINTS

# 6.1 Efficacy and Pharmacodynamic Endpoints

#### 6.1.1 Primary Efficacy Endpoint

• Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline at Week 4

# 6.1.2 Secondary Efficacy and Pharmacodynamic Endpoints

The key secondary endpoints are as follows:

- Absolute change in ppFEV<sub>1</sub> from baseline through Week 24
- Number of pulmonary exacerbations (PEx) through Week 24
- Absolute change in sweat chloride (SwCl) from baseline through Week 24
- Absolute change in Cystic Fibrosis Questionnaire Revised (CFQ-R) respiratory domain score from baseline through Week 24
- Absolute change in body mass index (BMI) from baseline at Week 24
- Absolute change in SwCl from baseline at Week 4
- Absolute change in CFQ-R respiratory domain score from baseline at Week 4

Other secondary endpoints

- Time-to-first PEx through Week 24
- Absolute change in BMI z-score from baseline at Week 24 (for subjects ≤20 years of age at Baseline)
- Absolute change in body weight from baseline at Week 24

#### 6.2 Safety Endpoints

Safety and tolerability will be evaluated via the following endpoints:

- Adverse events (AEs)
- Clinical laboratory values
- Standard 12-lead ECGs
- Vital signs
- Pulse oximetry

# 6.3 Pharmacokinetic Endpoint

• PK parameters of VX-445, TEZ, M1-TEZ, and IVA



#### 7 STUDY DESIGN

# 7.1 Overall Design

This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter study. A schematic of the study design is shown in Figure 7-1.

Figure 7-1 Schematic of the Study Design



IVA: ivacaftor; N: number of subjects; TEZ: tezacaftor

Notes: The figure is not drawn to scale. The Safety Follow-up Visit is not required for subjects who complete the Week 24 Visit and enroll in an open-label study within 28 days after the last dose of study drug (Section 9.1.3 of protocol).

Approximately 360 subjects will be randomized (1:1) to the VX-445/TEZ/IVA arm or the triple placebo arm. The planned dosages to be evaluated are shown in Table 7-1. Randomization will be stratified; details are provided in Section 9.2 of the CSP.

Table 7-1 Treatment Arms and Planned Dosages

| Treatment Arm | VX-445 Dosage | TEZ Dosage | IVA Dosage |
|---|---|---|---|
| VX-445/TEZ/IVA | 200 mg qd | $100 \mathrm{\ mg} \mathrm{\ qd}$ | 150 mg q12h |
| Triple placebo | $0~\mathrm{mg}$ | 0 mg | 0 mg |

IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TEZ: tezacaftor

Study visits and assessments to be conducted are shown in Section 3 of CSP. All visits will occur within the windows specified.

# 7.2 Sample Size and Power

Approximately 360 subjects will be enrolled and randomized (1:1) to the VX-445/TEZ/IVA arm or the triple placebo arm. This sample size was determined to provide adequate power for the key secondary endpoint of the number of PEx through Week 24. Information regarding the powering of primary and selected key secondary endpoints is provided below.

#### **Power for Primary Efficacy Endpoint**

The primary efficacy endpoint is the absolute change in ppFEV<sub>1</sub> from baseline at Week 4. The primary null hypothesis to be tested is that the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4 is the same for the 2 treatment groups, VX-445/TEZ/IVA and placebo. If the number of subjects included in the IA is 140, the null hypothesis will be tested at a 2-sided significance level of 0.044 during the IA and at an overall 2-sided significance level of 0.05. See Section 7.5 for details on the significance level for hypothesis testing during the IA.

Assuming a within-group SD of 7 percentage points and a 5% dropout rate at Week 4, an IA sample size of 70 subjects in each treatment group will have approximately 98% power to detect a difference between the treatment groups of 5.0 percentage points for the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4, based on a 2-sided, 2-sample t-test at a significance level of 0.044. If the P value fails to cross the efficacy boundary during the IA (P value  $\geq$ 0.044; assuming 140 subjects included in the IA), the primary endpoint of absolute change in ppFEV<sub>1</sub> from baseline at Week 4 will be tested after all subjects complete study participation at an alpha of 0.01. Assuming a 10% dropout rate at Week 24, a final analysis sample size of 180 subjects in each treatment group will have approximately 99% power to detect a difference between the treatment groups of 5.0 percentage points for the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4, based on a 2-sided, 2-sample t-test at a significance level of 0.01.

#### **Power for Selected Secondary Endpoints**

A key secondary endpoint is the absolute change in ppFEV<sub>1</sub> from baseline through Week 24. Assuming a within-group SD of 7 percentage points and a 10% dropout rate at Week 24, a sample size of 180 subjects in each treatment group will have approximately 99% power to detect a difference between the treatment groups of 5.0 percentage points for the absolute change in ppFEV<sub>1</sub> from baseline through Week 24, based on a 2-sided, 2-sample t-test at a significance level of 0.05.

A key secondary endpoint is the number of PEx through Week 24. Assuming a rate of PEx for the placebo group of 0.6 over 24 weeks and a 10% dropout rate, with 180 subjects and the overdispersion parameter of 0.5 in each treatment group, the power to detect a 40% reduction in the PEx rate for VX-445/TEZ/IVA group compared to placebo group is approximately 80%, based on a 2-sided, 2-sample negative binomial regression model test for the ratio of rates, at a significance level of 0.05.

#### 7.3 Randomization

Subjects will be randomized (1:1) to the VX-445/TEZ/IVA arm or to the triple placebo arm. Randomization will be stratified by ppFEV<sub>1</sub> determined during the Screening Period (<70 versus  $\ge 70$ ), age at the Screening Visit (<18 versus  $\ge 18$  years of age), and sex (male versus female).

An interactive web response system (IWRS) will be used to assign subjects to treatment. The randomization code list will be produced by Vertex Biometrics or a qualified randomization vendor.

Randomization will occur before the first dose of study drug during the Treatment Period and may occur on either Day 1 or Day -1.

# 7.4 Blinding and Unblinding

Refer to Section 10.7 of the CSP for details.

# 7.5 Interim Analysis

An IA is planned when at least 140 subjects complete the Week 4 Visit and at least 100 subjects complete the Week 12 Visit. The IA will be performed by an external independent biostatistician who is not involved in and will not influence the conduct of the study, and the results will be reviewed by an independent data monitoring committee (DMC). A Lan and DeMets<sup>3</sup> alpha spending function will be applied to control the overall type I error rate of 0.05 for the primary endpoints during the IA and the final analysis such that an alpha of 0.01 will be preserved for the final analysis. If the number of subjects included in the IA is 140, then the primary endpoint of the absolute change from baseline in ppFEV<sub>1</sub> at Week 4 will be tested at a significance level of 0.044 during the IA. The actual alpha at the IA ( $\alpha_0$ ) will be determined based on the actual number of subjects included in the interim Full Analysis Set (see Section 8.4.1).

Table 7-2 lists the actual alpha that will be spent at the IA with various numbers of subjects included in the interim Full Analysis Set. The actual number N along with the  $\alpha_0$  will be communicated to the independent biostatistician and DMC approximately 5 days prior to the IA data cut date.

Table 7-2 The Alpha Spending with Various N at the Interim Analysis

| Sample Size in interim Full Analysis Set (information fraction) | Alpha at IA $(\alpha_0)$ | Alpha at Final $(\alpha_1)$ |
|---|---|---|
| 140 (39%) | 0.0440 | 0.01 |
| 180 (50%) | 0.0451 | 0.01 |
| 220 (61%) | 0.0465 | 0.01 |
| 260 (72%) | 0.0480 | 0.01 |
| 300 (83%) | 0.0492 | 0.01 |

If the P value for the primary endpoint at the IA is less than  $\alpha_0$ , then the efficacy boundary has been crossed. If the DMC declares that the study has crossed the efficacy boundary, then the study may be unblinded to a limited Vertex team to prepare regulatory submission(s). Members of the limited Vertex unblinded team will not be involved in or influence the conduct of the remaining part of the study to protect the integrity of the study.

If the P value fails to cross the efficacy boundary during the IA (i.e., P value >=  $\alpha_0$ ), then the primary endpoint of absolute change in ppFEV<sub>1</sub> from baseline at Week 4 will be tested after all subjects complete study participation at an alpha of 0.01.

Selected key secondary endpoints will be analyzed during the IA with nominal P value provided for descriptive purpose (see Section 10.1.3.2).

#### 8 ANALYSIS SETS

#### 8.1 All Subjects Set

The **All Subjects Set** will include all subjects who are randomized or receive at least 1 dose of study drug. This analysis set will be used for all individual subject data listings and disposition summary tables, unless otherwise specified.

# 8.2 Full Analysis Set

The **Full Analysis Set** (FAS) will include all randomized subjects who carry the intended CFTR allele mutation and receive at least 1 dose of study drug. The FAS will be used to summarize subject demographics, baseline characteristics, and for all efficacy analyses in which subjects will be analyzed according to their randomized treatment group, unless otherwise specified.

# 8.3 Safety Set

The **Safety Set** will include all subjects who receive at least 1 dose of study drug. The Safety Set will be used for all safety analyses in which subjects will be analyzed according to the treatment they received, unless otherwise specified.

# 8.4 Analysis Sets for IA

A data cutoff date will be established for the IA as the latter of at least 140 subjects complete Week 4 Visit and at least 100 subjects complete Week 12 Visit.

All subjects randomized or dosed prior to the data cutoff date will be in the scope of the IA. All data reported on or before the data cutoff date will be included in the IA.

# 8.4.1 Interim Full Analysis Set

The **interim Full Analysis Set** (iFAS) will include subjects in the FAS whose scheduled Week 4 Visit is on or before the data cutoff date. That is, the iFAS will include subjects in the FAS who complete the Week 4 Visit or are randomized at least 28 days before the data cutoff date.

The iFAS will be used during the IA for subject demographics, baseline characteristics, and all efficacy analyses in which subjects will be analyzed according to their randomized treatment group.

# 8.4.2 Interim Safety Set

The **interim Safety Set** (IA Safety Set) will include subjects in the Safety Set who complete the Week 4 Visit or receive their first dose of study drug at least 28 days before the data cutoff date.

The IA Safety Set will be used during the IA for safety analyses in which subjects will be analyzed according to the treatment they received.

#### 9 STATISTICAL ANALYSIS

This section discusses the analyses planned for the final analysis. See Section 10.1 for the analyses planned for the IA.

#### 9.1 General Considerations

The Schedule of Assessments is provided in Section 3 of CSP. The precision standards for reporting safety and efficacy variables are provided in an internal Biometrics document that specifies the programming rules including the precision for derived variables.

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, SD, median, minimum value (min), and maximum value (max).

**Categorical variables** will be summarized using counts and percentages. Percentages will be presented to 1 decimal place.

**Baseline value**, unless otherwise specified, is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the Treatment Period.

**Absolute change** from baseline will be calculated as post-baseline value - baseline value.

**Relative change** from baseline will be calculated as (post-baseline value - baseline value)/baseline value.

**Treatment-emergent (TE) period** will include the time from the first dose of study drug in the Treatment Period until 28 days after the last dose of study drug or to the completion of study participation, whichever occurs first.

**Unscheduled visits:** Unscheduled visit measurements will be included in analysis as follows:

- 1) In scheduled visit windows per specified visit windowing rules
- 2) In the derivation of baseline and last on-treatment measurements
- 3) In the derivation of maximum and minimum values during TE period, and maximum and minimum change from baseline values during TE period for safety analyses
- 4) In individual subject data listings as appropriate

**Visit windowing rules:** The analysis visit windows for protocol-defined visits are provided in Appendix A.

**Incomplete/missing data** will not be imputed, unless otherwise specified.

**Outliers:** No formal statistical analyses will be performed to detect or remedy the presence of statistical outliers, unless otherwise specified.

#### 9.2 Background Characteristics

# 9.2.1 Subject Disposition

The number of subjects in the following categories will be summarized:

- All Subjects Set
- Full Analysis Set
- Safety Set
- Randomized
- Randomized but not dosed

The number and percentage (based on the FAS) of subjects in each of the following disposition categories will be summarized by treatment group and overall:

- Completed treatment
- Prematurely discontinued treatment and the reason for discontinuation
- Completed study
- Prematurely discontinued the study and the reason for discontinuation
- Rollover to open-label study

A listing will be provided for subjects who discontinued treatment or who discontinued study with reasons for discontinuation.

# 9.2.2 Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized by treatment group and overall based on the FAS.

Demographic data will include the following:

- Age at baseline (in years)
- Sex (male, female)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, and not collected per local regulations)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Other, and not collected per local regulations)
- Geographic region (North America, Europe [including Australia])

Baseline characteristics will include the following:

- Weight (kg)
- Height (cm)
- BMI  $(kg/m^2)$
- BMI z-score (for subjects ≤20 years old at Baseline)

Stratification categories (in addition to sex) will include the following:

- Age at the Screening Visit (<18, and  $\ge18$  years)
- ppFEV<sub>1</sub> determined during the Screening Period (<70, and  $\ge70$ )

Disease characteristics will include the following:

- ppFEV<sub>1</sub> at baseline ( $<40, \ge 40 \text{ to } <70, \ge 70 \text{ to } \le 90, \text{ and } >90$ )
- ppFEV<sub>1</sub> at baseline (continuous)
- Sweat chloride at baseline (continuous)
- CFQ-R respiratory domain score at baseline (continuous)
- Prior use of dornase alfa (Yes, No)
- Prior use of azithromycin (Yes, No)
- Prior use of inhaled antibiotic (Yes, No)
- Prior use of any bronchodilator (Yes, No)
- Prior use of any inhaled bronchodilator (Yes, No)
- Prior use of any inhaled hypertonic saline (Yes, No)
- Prior use of any inhaled corticosteroids (Yes, No)

• Infection with *Pseudomonas aeruginosa* within 2 years prior to screening (Positive, Negative)

In addition, data listings will also be provided for:

- Informed consent;
- Inclusion/Exclusion criteria violation for subjects with any such violations.

## 9.2.3 Medical History

Medical history will be coded by using the Medical Dictionary for Regulatory Activities (MedDRA). For the FAS, medical history will be summarized descriptively by system organ class (SOC) and preferred term (PT). The corresponding data listing will also be provided.

In addition, the number of subjects reported to have had positive cultures for respiratory pathogens within the 2 years prior to screening (i.e., answered yes on the respiratory microbiology form) will be summarized for the FAS. The corresponding data listing will be provided. Hospitalization and clinic visit history in the year prior to the signing of informed consent will be listed.

#### 9.2.4 Prior and Concomitant Medications

Medications will be coded using the World Health Organization Drug Dictionary (WHO-DD) and categorized as follows:

**Prior medication:** any medication that was administered during the 56 days before the first dose of study drug.

Concomitant medication: medication continued or newly received during the TE period.

**Post-treatment medication:** medication continued or newly received after the TE period.

A given medication may be classified as follows: prior, concomitant, post-treatment, both prior and concomitant, both concomitant and post-treatment, or prior, concomitant, and post-treatment.

If a medication has a completely missing or partially missing start/stop date and it cannot be determined whether it was taken before the first dose date of study drug, concomitantly during the TE period, or after the TE period, it will be classified as prior, concomitant, and post-treatment.

For the FAS, prior medications and concomitant medications will be summarized descriptively by: 1) treatment group and overall, preferred name (PN); and 2) treatment group and overall, anatomic class (ATC) level 1, ATC level 2, and PN. Post-treatment medications will be listed for each subject.

Details for imputing missing or partial start and/or stop dates of medication are described in Appendix B.

# 9.2.5 Study Drug Exposure

Duration of study drug exposure (in days) will be calculated as: last dose date of study drug – first dose date of study drug + 1, regardless of study drug interruption.

Study drug exposure (in weeks) will be summarized descriptively by the number of subjects (n), mean, SD, median, min, and max. It will also be summarized in categories for Treatment Period:  $\leq 1$  weeks,  $\geq 1-\leq 2$  weeks,  $\geq 2-\leq 4$  weeks,  $\geq 4-\leq 8$  weeks,  $\geq 8-\leq 12$  weeks,  $\geq 12-\leq 16$  weeks,  $\geq 16-\leq 20$  weeks,  $\geq 20-\leq 24$  weeks, and  $\geq 24$  weeks, using counts and percentages. Additionally, the total study drug exposure, defined as the sum total of the study drug exposure across all subjects (in patient-weeks and patient-years), will be provided.

Exposure summaries will be based on the Safety Set, and presented by treatment group and overall.

# 9.2.6 Study Drug Compliance

Study drug compliance will be calculated as:  $100 \times [1 - (total number of days of study drug interruption) / (duration of study drug exposure in days)]. A study drug interruption on a given day is defined as an interruption of any study drug on that day. A study drug interruption that continues through the end of the study participation (i.e., subject does not resume study drug before the end of the study participation) will not be included in the compliance calculation.$ 

Percentage of study drug compliance will be summarized based on the FAS, and presented by treatment group and overall. Percentage of study drug compliance will be summarized descriptively by the number of subjects (n), mean, SD, median, min, and max. It will also be summarized in categories: <80% and  $\ge80\%$  using frequency tables.

In addition, percentage of tablets taken will be calculated using the following formula:  $100 \times [(\text{total number of tablets dispensed}) - (\text{total number of tablets returned})] / (\text{total number of tablets planned to be taken per day} \times \text{duration of study drug exposure in days}). Summary similar to those for the study drug compliance will be produced based on the FAS.$ 

# 9.2.7 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. IPD rules will be developed and finalized prior to the IA data lock.

The protocol deviations that should be considered as potential IPDs include, but are not limited to:

- Subject was enrolled in the study despite the violation of inclusion/exclusion criteria
- Subject was less than 80% compliant with study drug for non-safety reason
- Subject received prohibited concomitant medications
- Subject received the wrong treatment or incorrect doses
- Subject remained in the study despite meeting withdrawal criteria

Occurrence of any of these events should be considered as potential IPDs, but a blinded team should categorize them as IPDs only if they have the potential to significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being.

IPDs (from the clinical database or from the site deviation log) will be summarized descriptively based on the FAS and presented by treatment group and overall. Additionally, IPDs will be provided in an individual subject data listing.

# 9.3 Efficacy Analysis

All efficacy analyses described in this section will be based on the FAS, unless otherwise specified.

#### 9.3.1 Analysis of Primary Efficacy Variable

#### 9.3.1.1 Definition of Variables

The primary efficacy variable is the absolute change in  $ppFEV_1$  from baseline at Week 4. Percent predicted  $FEV_1$  is the ratio of  $FEV_1$  (L) and predicted  $FEV_1$  (L), expressed as a percentage. See Appendix C for more details.

# 9.3.1.2 Primary Analysis

The primary analysis will be performed using a mixed-effects model for repeated measures (MMRM) with change from baseline at Day 15, Week 4, Week 8, Week 12, Week 16, and Week 24 as the dependent variable. The model will include treatment group, visit, and treatment by visit interaction as fixed effects, with continuous baseline ppFEV<sub>1</sub>, age at screening (<18 versus  $\ge$ 18 years of age) and sex (male versus female) as covariates. The model will be estimated using restricted maximum likelihood. Denominator degrees of freedom for the *F*-test for fixed effects will be estimated using the Kenward-Roger approximation<sup>2</sup>. An unstructured covariance structure will be used to model the within-subject errors. If the model estimation does not converge, a compound symmetry covariance structure will be used instead. Conditional on the observed data and covariates, missing data will be assumed to be missing at random; consequently, no imputation of missing data will be performed.

The primary result obtained from the model will be the estimated treatment difference at Week 4. The adjusted means with 2-sided 95% confidence intervals and 2-sided *P* values will be provided. Furthermore, the treatment difference at each post-baseline visit obtained from the model will also be provided.

# 9.3.1.3 Supportive Analyses

There will be no supportive analysis for the primary efficacy endpoint.

#### 9.3.1.4 Sensitivity Analyses

#### MMRM based on Multiple Imputation (MI)

An underlying assumption of the MMRM method is that data are missing at random. To minimize the amount of missing data, subjects who prematurely discontinue study drug treatment will continue to complete all scheduled study visits for spirometry and other efficacy assessments.

To assess the impact of missing data and the assumption that data are missing at random, a multiple imputation algorithm will be used if  $\geq 10\%$  of the subjects have missing change in ppFEV<sub>1</sub> at Week 24 in any treatment group. Missing absolute change from baseline in ppFEV<sub>1</sub> assessments will be imputed starting from the first visit with missing values, for which all subsequent visits through Week 24 are also missing. For intermediate missing data, i.e., missing values that fall between two non-missing ones, it is reasonable to assume that they are missing at

random and therefore will not be imputed. An MMRM analogous to that for the primary analysis of the primary endpoint will be applied to imputed datasets and the relevant MI estimators will be reported. Details for the MI steps are presented in Appendix D.

# 9.3.1.5 Subgroup Analysis

Subgroup analyses of the primary efficacy endpoint will be performed using a model similar to that of the primary analysis for each of the following subgroups:

- Age at screening ( $<18, \ge 18$  years)
- Percent predicted FEV<sub>1</sub> at baseline ( $<70, \ge 70$ )
- Sex (male, female)
- Geographic region (North America, Europe [including Australia])
- Prior use of inhaled antibiotic (Yes, No)
- Prior use of dornase alfa (Yes, No)
- Prior use of inhaled bronchodilator (Yes, No)
- Prior use of inhaled hypertonic saline (Yes, No)
- Prior use of inhaled corticosteroids (Yes, No)
- Prior use of azithromycin (Yes, No)
- Infection with *Pseudomonas aeruginosa* within 2 years prior to screening (Positive, Negative)

The MMRM used for the primary analysis will be used for the subgroup analysis, where the same model will be applied to each category of the subgroup. Note that for the subgroup analysis based on age and sex, the covariate of age at screening (<18 versus ≥18 years of age) and sex (male versus female) from the MMRM will be removed, respectively. The adjusted means with 2-sided 95% confidence intervals will be provided. Furthermore, the estimated treatment difference at Week 4 in different categories within a subgroup will also be presented in a forest plot. Note: The results from the subgroup analysis should be interpreted with caution in the cases where sample sizes are small.

# 9.3.2 Analysis of Key Secondary Variables

#### 9.3.2.1 Definition of Variables

<u>Pulmonary exacerbation (PEx)</u>: A PEx is defined as a new event or change in antibiotic therapy (IV, inhaled, or oral) for any 4 or more of the following signs/symptoms:

- Change in sputum
- New or increased hemoptysis
- Increased cough
- Increased dyspnea
- Malaise, fatigue, or lethargy

- Temperature above 38°C (equivalent to approximately 100.4°F)
- Anorexia or weight loss
- Sinus pain or tenderness
- Change in sinus discharge
- Change in physical examination (PE) of the chest
- Decrease in pulmonary function by 10%
- Radiographic changes indicative of pulmonary infection

The **PEx analysis period** will include the time from the first dose date of study drug until the last efficacy assessment, which may be collected up to the Week 24 Visit or the earlier of Day 169 and the end of study participation if subject does not have the Week 24 Visit.

The number of PEx through Week 24 is then defined as the total number of PEx for each treatment group during the PEx analysis period.

Sweat chloride (SwCl): the SwCl value for a given visit will be calculated as the mean of the non-missing sweat chloride measurements obtained on the left and right arms at that visit. If one of the two arm measurements at a time point is missing, the other will be used as the mean. A volume  $\geq 15~\mu L$  is required for an accurate determination of sweat chloride. Any results reported as having volume  $<15~\mu L$  will be considered missing. Any sweat chloride values reported as <10~mmol/L or >160~mmol/L will be considered missing.

<u>Cystic Fibrosis Questionnaire-Revised (CFQ-R)</u>: The CFQ-R<sup>1,4,6</sup> is a validated CF-specific instrument that measures quality-of-life domains. This study utilizes three different versions of CFQ-R:

- CFQ-R for Children ages 12 and 13
- CFQ-R for Adolescents and Adults (subjects 14 years and older)
- CFQ-R for Parents/Caregivers (subjects 13 years and younger)

In all three versions, specific question belonging to a domain is scored 1, 2, 3, or 4. The CFQ-R domain score, e.g., physical domain score or respiratory domain score, is defined as a scaled score as follows:

Scaled score for a domain =  $100 \times (\text{mean (scores of all questions in the domain)} - 1)/3,$ 

where the score from a negatively phrased question is first reversed, i.e., reversed score = 5 – actual score, so that 1 always represents the worst condition and 4 the best condition. The (scaled) domain score ranges from 0 (worst condition) to 100 (best condition). The scaled score for a specific domain will not be calculated if more than half of the questions in the domain have missing scores.

The (scaled) domain score from the CFQ-R for Children ages 12 and 13 and for Adolescent and Adults will be pooled for the analysis purpose.

<u>Body mass index (BMI)</u>: the BMI at each visit is calculated using the weight and height at each visit as follows:

$$BMI = \frac{Weight (kg)}{Height (m^2)}$$

# 9.3.2.2 Analysis Method

Absolute change in  $ppFEV_1$  through Week 24: Analysis of this variable will be based on an MMRM that is exactly the same as the primary efficacy variable. However, the Day 15 Visit will not be included in the estimation of the average treatment effect through Week 24 as the treatment effect is not expected to reach the steady state at Day 15.

Number of PEx through Week 24: Analysis of this variable will be performed using a negative binomial regression model with a fixed effect for treatment, as well as continuous baseline ppFEV<sub>1</sub>, age at screening (<18 versus  $\ge18$  years of age), and sex (male versus female) as covariates. The logarithm of the subject-specific PEx analysis period duration (in years) will be treated as the offset in the model.

Absolute change in SwCl from baseline through Week 24: Analysis of this PD variable will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Week 4, Week 8, Week 12, and Week 24 Visits will be included in the model and all of these visits will be included in the estimation of the average treatment effect through Week 24.

Absolute change in the CFQ-R respiratory domain score from baseline through Week 24: Analysis of this domain will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Week 4, Week 8, Week 12, Week 16, and Week 24 Visits will be included in the model and all of these visits will be included in the estimation of the average treatment effect through Week 24.

Absolute change in BMI from baseline at Week 24: Analysis of this variable will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Day 15, Week 4, Week 8, Week 12, Week 16, and Week 24 Visits will be included in the model.

Absolute change in SwCl from baseline at Week 4: Analysis of this PD variable will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Week 4, Week 8, Week 12, and Week 24 Visits will be included in the model to estimate the treatment effect at Week 4.

Absolute change in CFQ-R respiratory domain score from baseline at Week 4: Analysis of this domain will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Week 4, Week 8, Week 12, Week 16 and Week 24 Visits will be included in the model to estimate the treatment effect at Week 4.

To assess the longitudinal profile of the efficacy and pharmacodynamic assessments with repeated measures up to Week 24, the LS mean (SE) of the within-treatment group change from baseline at each post-baseline visit along with the 95% CI will be estimated from the corresponding MMRM. The LS mean (SE) of the treatment difference between VX-445/TEZ/IVA and triple placebo at each post-baseline visit will be provided along with the corresponding 95% CI and *P* value. The LS mean (SE) at each visit will also be plotted by treatment group. In addition, the post-baseline raw values and the absolute change from baseline at each post-baseline visit will be summarized descriptively (n, mean, SD, median, minimum, and maximum).

# 9.3.2.3 Multiplicity Adjustment

The Lan and DeMets<sup>3</sup> alpha spending function will be applied to the primary endpoint of the absolute change in ppFEV<sub>1</sub> at Week 4 to control the overall type I error rate of 0.05 such that an alpha of 0.01 will be preserved for the final analysis.

If the number of subjects included in the IA is 140, the primary endpoint of the absolute change from baseline in ppFEV<sub>1</sub> at Week 4 will be tested at an alpha of 0.044 during the IA. The actual alpha at the IA ( $\alpha_0$ ) will be determined based on the actual number of subjects included in the interim Full Analysis Set. If the study does not cross the efficacy boundary during the IA (P value  $\geq \alpha_0$ ), then the primary endpoint will be tested at an alpha of 0.01 at the final analysis when all subjects complete the study participation. See Section 7.5 for more details.

The key secondary endpoints will be formally tested at an alpha of 0.05 at the final analysis when all subjects complete study participation only if the primary endpoint is statistically significant at the IA or at the final analysis. A hierarchical testing procedure will be used to control the type I error rate for the multiple key secondary endpoints tested at an alpha of 0.05. For a test at any step to be considered statistically significant within the testing hierarchy, it must be statistically significant, and all previous tests (if any) within the hierarchy must be statistically significant at the 0.05 level. The testing order of the key secondary endpoints is as follows:

- Absolute change in ppFEV<sub>1</sub> from baseline through Week 24
- Number of PEx through Week 24
- Absolute change in SwCl from baseline through Week 24
- Absolute change in CFQ-R respiratory domain from baseline through Week 24
- Absolute change in BMI from baseline at Week 24
- Absolute change in SwCl from baseline at Week 4
- Absolute change in CFQ-R respiratory domain score from baseline at Week 4

# 9.3.3 Analysis of Other Secondary Variables

#### 9.3.3.1 Definition of Variables

<u>Time-to-first PEx through Week 24</u>: the number of days from the first dose date of study drug to the date of the first pulmonary exacerbation during the PEx analysis period. A subject who does not experience a PEx during the PEx analysis period will be censored at the PEx analysis period end date.

<u>BMI z-score</u>: the BMI score, adjusted for age and sex, will be referred to as BMI-for-age z-score (BMI z-score). The BMI z-score will be calculated by using Centers for Disease Control and Prevention (CDC) growth charts<sup>8</sup>, with the age (in months) used for the calculation defined in Appendix A.

# 9.3.3.2 Analysis Method

<u>Time-to-first PEx through Week 24</u>: Time-to-first PEx will be analyzed using the Cox regression model. The model will include a fixed effect for treatment, as well as continuous baseline ppFEV<sub>1</sub>, age at screening (<18 versus  $\ge18$  years of age), and sex (male versus female) as

covariates. Additionally, the Kaplan-Meier method will be used to estimate the cumulative exacerbation-free rate by treatment group; the associated plot will be provided.

Note: If the number of events is <5 in either treatment group, Cox regression will not be performed and the analysis of the time-to-first PEx will be restricted to the Kaplan-Meier method.

Absolute change in BMI z-score from baseline at Week 24 (for subjects ≤20 years of age at Baseline): Analysis of this variable will be based on an MMRM similar to the analysis of the primary efficacy variable, excluding the covariate of age at screening (<18 versus ≥18 years of age), for subjects ≤20 years of age at Baseline. Data obtained from Day 15, Week 4, Week 8, Week 12, Week 16, and Week 24 Visits will be included in the model.

Absolute change in body weight from baseline at Week 24: Analysis of this variable will be based on an MMRM similar to the analysis of the primary efficacy variable. Data obtained from Day 15, Week 4, Week 8, Week 12, Week 16, and Week 24 Visits will be included in the model.





# 9.3.4.3 Analysis of Additional Variables for Pulmonary Exacerbations and Hospitalization

The analysis period for all variables in this section will be the same as the PEx analysis period.

# **Pulmonary Exacerbations**

In addition to the key secondary endpoints, PEx will be further analyzed as described below:

- Time-to-first event (time in days):
  - o Time-to-first PEx requiring hospitalization
  - o Time-to-first PEx requiring IV antibiotic therapy
  - o Time-to-first PEx requiring hospitalization or IV antibiotic therapy
- Number of events
  - Number of PEx requiring hospitalizations
  - o Number of PEx requiring IV antibiotic therapy
  - o Number of PEx requiring hospitalization or IV antibiotic therapy
- Duration of events:
  - Number of days with PEx
  - o Number of days with PEx requiring hospitalization
  - o Number of days with PEx requiring IV antibiotic therapy
  - o Number of days with PEx requiring hospitalization or IV antibiotic therapy.

#### Hospitalization

- Number of events:
  - o Number of planned hospitalizations for CF (i.e., antibiotic therapy)
  - Number of all unplanned hospitalizations for reasons other than antibiotic therapy for sinopulmonary signs/symptoms
- Duration of events
  - o Number of days of all unplanned hospitalizations for reasons other than antibiotic therapy for sinopulmonary signs/symptoms

For the time to event variables, the analysis time will be the number of days from the first dose date of study drug to the date of the first defined event during the PEx analysis period. A subject who does not experience the event during the PEx analysis period will be censored at the PEx analysis period end date for that event.

For the number of events variables, subjects with multiple defined events during the PEx analysis period will be counted multiple times. The annualized duration of events for each subject will be the total number of days with the defined events times 48 weeks divided by the total number of weeks on study up to the end of the PEx analysis period.

# Analysis of Pulmonary/Hospitalization Variables

**Time-to-first event**: the time-to-first event endpoints will be analyzed similarly to the analysis of time-to-first PEx described in Section 9.3.3.2.

Note: If the number of subjects with events is <5 in either treatment group, Cox regression will not be performed and analysis of time-to-first event will be restricted to Kaplan-Meier methods.

**Number of events**: the number of events will be analyzed using negative binomial regression similar to the analysis of number of PEx described in Section 9.3.2.2.

Note: If the number of events is <5 in either treatment group, negative binomial regression will not be performed and analysis of event counts will be based on a Fisher's Exact test.

**Duration (number of days)**: the annualized duration of events will be analyzed using a stratified (by ppFEV<sub>1</sub> at screening (<70 versus  $\ge$ 70), age at screening (<18 versus  $\ge$ 18 years of age), and sex (male versus female)) Wilcoxon rank-sum test to assess the difference between treatment groups.

# 9.4 Safety Analysis

All safety analyses will be based on data from the TE period for all subjects in the Safety Set. Subjects will be analyzed according to the treatment they actually received in the Treatment Period. For subjects receiving study drug from more than one treatment group, the treatment group allocation will be the higher treatment group (VX-445/TEZ/IVA > TC Placebo).

The overall safety profile of the study drug will be assessed in terms of the following safety and tolerability endpoints:

- Treatment-emergent adverse events (TEAEs)
- Clinical laboratory values
- ECGs
- Vital signs
- Pulse oximetry

Only descriptive analysis of safety will be performed and no statistical testing will be performed.

#### 9.4.1 Adverse Events

For analysis purposes, AEs will be classified as pretreatment AEs, TEAEs, or post-treatment AEs, defined as follows:

**Pretreatment AE:** any AE that occurred before the first dose date of study drug

**TEAE:** any AE that worsened (either in severity or seriousness) or that was newly developed at or after the first dose date of study drug through the end of the TE period

**Post-treatment AE:** any AE that worsened (either in severity or seriousness) or that was newly developed after the TE period

For AEs with completely missing or partially missing start dates, if there is no clear evidence that the AEs are pre-treatment or post-treatment, the AEs will be classified as TEAEs.

Details for imputing missing or partial start dates of adverse events are described in Appendix E.

An overview of all TEAEs by treatment group and overall will be summarized in the following categories:

- Number of TEAEs (total number of TEAEs only)
- Subjects with any TEAEs
- Subjects with TEAEs by strongest relationship
- Subjects with TEAEs by maximum severity
- Subjects with TEAEs leading to study drug discontinuation (discontinuation of any study drug)
- Subjects with TEAEs leading to study drug interruption (interruption of any study drug)
- Subjects with Grade 3/4 TEAEs
- Subjects with related TEAEs
- Subjects with serious TEAEs
- Subjects with related serious TEAEs
- Subjects with TEAE leading to death

The following summary tables of TEAEs will be presented by treatment group:

- All TEAEs
- Grade 3/4 TEAEs
- TEAEs by strongest relationship
- TEAEs by maximum severity
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- Related TEAEs
- Serious TEAEs
- Related serious TEAEs
- TEAEs leading to death

Summaries will be presented by MedDRA SOC and PT using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentages of subjects, subjects with multiple occurrences of the same adverse event or a continuing adverse event will be counted once, and only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries.

Additional summary tables will be presented by treatment for TEAEs showing number and percentage of subjects

# • All TEAEs by PT

All AEs, including pretreatment AEs, TEAEs, and post-treatment AEs, will be presented in an individual subject data listing based on the All Subjects Set. In addition, a listing containing individual subject adverse event data for TEAEs leading to treatment discontinuation, TEAEs leading to treatment interruption, Grade 3/4 TEAEs, SAEs and all deaths will be provided separately, with a flag indicating the TEAE status for SAEs and deaths.

For all AEs, the eCRF captures the action taken for VX-445/TEZ/IVA pills separately from the action taken for IVA monotherapy pills. As a result, it is possible that, in the final database (after database lock), the AE actions taken for the two agents (fixed dose VX-445/TEZ/IVA and ivacaftor monotherapy) are different. The summaries and listings of "AE Leading to Treatment Dis continuation" and "AE Leading to Treatment Interruption" account for discontinuation and interruptions for either agent.

#### 9.4.1.1 Subgroup Analysis

An overview of all TEAEs and a summary of TEAEs by SOC and PT for the following subgroups will be provided:

- Age at screening ( $<18, \ge 18$  years)
- Percent predicted FEV<sub>1</sub> at baseline ( $<70, \ge 70$ )
- Sex (male, female)
- Geographic Region (North America, Europe [including Australia])

# 9.4.2 Clinical Laboratory

For the treatment-emergent laboratory assessments, the observed values and change from baseline values of the continuous hematology, coagulation and chemistry results will be summarized in SI units at each visit by treatment group.

The number and percentage of subjects meeting at least 1 threshold analysis criterion event during the TE period will be summarized by treatment group. The threshold analysis criterion shift from baseline will also be summarized for selected laboratory parameters. The threshold analysis criteria are provided in Appendix F.

For select LFT laboratory tests (alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase [ALP], and total bilirubin), a scatter plot of the maximum treatment-emergent value versus the baseline value corresponding to ×ULN (upper limit of normal) will be presented. Further, a scatter plot of the maximum treatment-emergent value of ALT and AST,

separately, versus the maximum treatment-emergent value of total bilirubin corresponding to ×ULN will also be presented by treatment group.

Results of positive urine/serum pregnancy test will be listed in individual subject data listings only. For positive serum pregnancy listing, subjects with serum HCG which are abnormally high will be selected.

In addition, a listing containing individual subject hematology, chemistry, and coagulation values will be provided. This listing will include data from both scheduled and unscheduled visits.

# 9.4.3 Electrocardiogram

For the treatment-emergent ECG measurements, a summary of observed values and change from baseline values will be provided at each visit by treatment group for the following ECG measurements (in msec): RR interval, PR interval, QT interval, and QTcF interval, QRS duration, and Heart Rate (beats per minute).

The number and percentage of subjects meeting at least 1 threshold analysis criterion during the TE period will be summarized by treatment group. The threshold analysis criteria are provided in Appendix F.

#### 9.4.4 Vital Signs

For the treatment-emergent vital signs measurements, the observed values and change from baseline values will be summarized at each visit by treatment group. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

The number and percentage of subjects meeting at least 1 threshold analysis criterion during the TE period will be summarized by treatment group. The threshold analysis criteria are provided in Appendix F.

#### 9.4.5 Pulse Oximetry

For the treatment-emergent pulse oximetry measurements, a summary of observed values and change from baseline values will be provided at each visit by treatment group, for the percent of oxygen saturation by pulse oximetry.

The number and percentage of subjects with shift changes from baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the TE period will be summarized by treatment group.

#### 9.4.6 Physical Examination

Abnormal PE findings will be presented as an individual subject data listing only.

# 9.4.7 Supportive Safety Analysis

#### 9.4.7.1 Adverse Events of Special Interest

For this study, elevated transaminase events and rash events, as determined by MedDRA preferred terms in Appendix G, are considered as adverse events of special interest.

For treatment-emergent elevated transaminase events and rash events, the following categories will be summarized by treatment group:

• Subjects with events

- Subjects with events by maximum severity
- Subjects with events leading to treatment discontinuation
- Subjects with events leading to treatment interruption
- Subjects with serious events
- Subjects with related serious events
- Subjects with events leading to death
- Duration of events
- Time-to-onset of first event

In addition, for treatment-emergent rash events, these categories will be summarized for the following subgroups:

- Sex (male, female)
- Female subjects with concomitant hormonal therapy (Yes, No)

# 9.4.7.2 Hormonal Therapy

The number of subjects who used hormonal therapy concomitantly will be summarized by treatment group based on the Safety Set.



#### 10 SUMMARY OF INTERIM AND DMC ANALYSIS

For each DMC meeting and the planned IA, the Vertex Biometrics Department will prepare the analysis package using the dummy treatment code and dummy spirometry and SwCl data according to the DMC charter and the DMC SAP, respectively; SAS (Version 9.4, or higher) will be used to generate all statistical outputs (tables, figures, listings, and datasets).

, appointed as the independent biostatistician, will perform the IA according to the DMC SAP using the SAS code provided by Vertex Biometrics Department, the unblinded treatment code, the real (restricted) spirometry, and the real (restricted) sweat chloride data. Unblinded treatment code, spirometry, and sweat chloride data will be transferred directly from relevant vendors to the independent biostatistician. will present the results to the DMC.

If the study crosses the efficacy boundary according to the pre-specified criterion (Section 7.5), a limited Vertex unblinded team may be unblinded to the study. The limited Vertex unblinded team will use the unblinded treatment code and real (restricted) data to generate statistical outputs and prepare for submission(s). Members of the limited Vertex unblinded team will not be involved in or influence the conduct of the remaining part of the study to protect the integrity of the study.

#### 10.1 Interim Analysis

# 10.1.1 General Consideration

Refer to Section 7.5 for the timing of the IA. General considerations, reporting conventions, and analysis methods specified for the final analysis apply to the IA, unless otherwise specified.

For the IA purpose, the **treatment-emergent (TE) period** will include the time from the first dose of study drug in the Treatment Period until 28 days after the last dose of study drug, or the study participation end date, or the IA data cutoff date, whichever occurs first.

# 10.1.2 Background Characteristics

#### 10.1.2.1 Subject Disposition

The number of subjects in the following categories will be summarized:

- All Subjects Set
- Interim Full Analysis Set
- IA Safety Set
- Safety Set
- Randomized
- Randomized but not dosed

The number and percentage (based on the iFAS) of subjects in each of the following disposition categories will be summarized by treatment group and overall:

- Completed Week 4 Visit
- Prematurely discontinued treatment before Week 4 Visit and the reason for discontinuation
- Completed Week 12 Visit
- Prematurely discontinued treatment before Week 12 Visit and the reason for discontinuation
- Completed treatment
- Prematurely discontinued treatment and the reason for discontinuation
- Completed study
- Prematurely discontinued the study and the reason for discontinuation
- Rollover to open-label study

A listing will be provided for subjects who discontinued treatment or who discontinued study with reasons for discontinuation.

# 10.1.2.2 Demographics and Baseline Characteristics

The same demographics and baseline characteristics specified in Section 9.2.2 will be summarized based on the iFAS.

# 10.1.2.3 Study Drug Exposure

For the purpose of the IA, the study drug exposure will be calculated using the same approach specified in Section 9.2.5. For subjects who are still on study drug at the IA data cutoff date, the IA data cutoff date will be used as the last dose date for the exposure calculation.

Exposure summaries will be provided for subjects in the IA Safety Set as well as for subjects in the Safety Set who had been on-study for  $\geq$ 12 weeks, and will be presented by treatment group and overall.

# 10.1.3 Efficacy Analysis

All efficacy analyses described in this section will be based on the iFAS, unless otherwise specified.

#### 10.1.3.1 Analysis of Primary Efficacy Variable

The analysis of the primary efficacy variable of absolute change in ppFEV<sub>1</sub> from baseline at Week 4 will be performed using an MMRM with change from baseline at Day 15 and Week 4 as the dependent variable. The model will include treatment group, visit, and treatment by visit interaction as fixed effects, with continuous baseline ppFEV<sub>1</sub>, age at screening (<18 versus  $\geq$ 18 years of age) and sex (male versus female) as covariates. The model will be estimated using restricted maximum likelihood. Denominator degrees of freedom for the *F*-test for fixed effects will be estimated using the Kenward-Roger approximation<sup>2</sup>. An unstructured covariance structure will be used to model the within-subject errors. If the model estimation does not converge, a compound symmetry covariance structure will be used instead. Conditional on the observed data and covariates, missing data will be assumed to be missing at random; consequently, no imputation of missing data will be performed.

The sensitivity analysis based on the multiple imputation (Section 9.3.1.4) will be performed during the IA, if  $\geq 10\%$  of the subjects have missing change in ppFEV<sub>1</sub> at Week 4 in any treatment group. However, since the analysis model uses the change from baseline at Day 15 and Week 4 as the dependent variable, the primary timepoint for imputation will be Week 4 and only data up to the Week 4 Visit will be used in the imputation.

Subgroup analyses of the primary efficacy variable will also be performed during the IA in a manner similar to that of the primary analysis (Section 9.3.1.5) for each of the following subgroups using data up to the Week 4 Visit:

- Age at screening ( $<18, \ge 18$  years)
- Percent predicted FEV<sub>1</sub> at baseline ( $<70, \ge 70$ )
- Sex (male, female)
- Geographic region (North America, Europe [including Australia])

# 10.1.3.2 Analysis of Key Secondary Efficacy Variable

The following key secondary efficacy variables defined in Section 9.3.2.1 will be analyzed during the IA using an ANCOVA model:

- Absolute change in SwCl from baseline at Week 4
- Absolute change in CFQ-R respiratory domain score from baseline at Week 4

The model will use the change from baseline value at Week 4 as the dependent variable and include treatment group as fixed effects with continuous baseline ppFEV<sub>1</sub>, age at screening (<18 versus  $\ge$ 18 years of age), and sex (male versus female) as covariates. The estimated treatment difference at Week 4, the adjusted means with 2-sided 95% confidence intervals and nominal 2-sided P values will be provided.

Analyses of other efficacy and/or pharmacodynamic variables may be performed if the data are deemed sufficient.

# 10.1.3.3 Summary of Efficacy Variables

The raw value and change from baseline in ppFEV<sub>1</sub>, SwCl and CFQ-R will be summarized descriptively (n, mean, SD, median, minimum, and maximum) at baseline and post-baseline visits. For the IA purpose, a visit will be included in the summary if there are  $\geq$ 20 subjects with available data from each treatment group at that visit.

# 10.1.4 Safety Analysis

Safety analyses specified in Section 9.4 will be performed during the IA based on the IA Safety Set.

# 10.1.4.1 Additional Safety Analysis

The following safety summaries will be performed during the IA based on the Safety Set, as well as for subjects in the Safety Set who had been on-study for  $\geq 12$  weeks.

- An overview of all TEAEs by treatment group and overall which includes the following categories:
  - o Number of TEAEs (total number of TEAEs only)

- Subjects with any TEAEs
- o Subjects with TEAEs by strongest relationship
- Subjects with TEAEs by maximum severity
- O Subjects with TEAEs leading to study drug discontinuation
- o Subjects with TEAEs leading to study drug interruption
- Subjects with Grade 3/4 TEAEs
- Subjects with related TEAEs
- Subjects with serious TEAEs
- Subjects with related serious TEAEs
- Subjects with TEAE leading to death
- Summaries of TEAEs by MedDRA SOC and PT using frequency counts and percentages, presented by treatment group, for the following:
  - o All TEAEs
  - o Grade 3/4 TEAEs
  - TEAEs leading to treatment discontinuation
  - o TEAEs leading to treatment interruption
  - Serious TEAEs
- A summary of TEAEs by PT
- Analysis of adverse events of special interest (see Section 9.4.7.1)
- Threshold analysis for the LFT laboratory test (see Section 9.4.2)

#### 10.2 DMC Analysis

The DMC will conduct planned safety/efficacy review(s) of study data as outlined in the DMC charter. For the open session of each DMC meeting, selected tables will be presented for the overall treatment group based on the blinded data. For the closed session, the presentation will be by treatment group based on the unblinded data (generated by the independent biostatistician).

The timing of DMC meetings is outlined in Table 10-1.

**Table 10-1 DMC Meeting Schedule** 

| Meeting | Timing |
|---|---|
| Organizational | Teleconference prior to start of the study |
| First Planned Review | After ≥50 subjects have completed Week 4 |
| Second Planned<br>Review | Interim analysis of safety and efficacy after $\geq$ 140 subjects have completed the Week 4 visit and after $\geq$ 100 subjects have completed the Week 12 visit. |
| Ad-hoc | Teleconference on an as-needed basis |

# 10.2.1 DMC Safety/Efficacy Review

To protect the integrity of the treatment assignment and study data, the following steps for the flow of data will be executed for the DMC review:

- 1. The Vertex Biometrics Department will prepare the SAS codes, SDTM/ADaM data sets, and blinded outputs (tables, figures and listings) of safety and efficacy data using dummy treatment codes, dummy (unrestricted) spirometry data, and dummy (unrestricted) sweat chloride data;
- 2. The IWRS vendor, will provide the unblinded treatment codes to the independent biostatistician via a secure file transfer protocol, the independent biostatistician will verify the treatment assignment against the randomization list generated by
- 3. The spirometry vendor will provide the restricted spirometry data directly to the independent biostatistician, via a secure file transfer protocol;
- 4. The sweat chloride vendor will provide the restricted sweat chloride data directly to independent biostatistician, via a secure file transfer protocol;
- 5. The independent biostatistician will generate the unblinded outputs (tables, figures and listings) and provide them directly to the DMC team for their review, via a secure file transfer protocol.
- 6. The Vertex Biometrics Department will generate any blinded outputs (tables, figures and listings), for the open sessions of the DMC meetings, as applicable.

#### 11 REFERENCES

- <sup>1</sup> Goss C, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac Soc. 2007;4:1-9.
- <sup>2</sup> Kenward MG, Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. Biometrics. 1997;53:983-97.
- <sup>3</sup> Lan KK, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika. 1983;70(3):445-63.
- <sup>4</sup> Modi AC, Quittner AL. Validation of a disease-specific measure of health-related quality of life for children with cystic fibrosis. J Pediatr Psychol. 2003;28(8):535-45.
- <sup>5</sup> Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall G, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.
- <sup>6</sup> Quittner AL, Modi A, Cruz I. Systematic review of health-related quality of life measure for children with respiratory conditions. Pediatr Respir Rev. 2008;9:220-32.
- <sup>7</sup>Rubin, DB. and Schenker, N.. Interval estimation from multiply-imputed data: a case study using agriculture industry codes. Journal of the American Statistical Association. 1987; 81: 366–374.
- <sup>8</sup> Centers for Disease Control and Prevention. CDC Growth Charts. Available at: http://www.cdc.gov/growthcharts/percentile data files.htm.

# 12 LIST OF APPENDICES

# Appendix A: Analysis Visit Windows for Safety and Efficacy Assessments

| Assessment | Visit <sup>1</sup> | Target Study Day | Analysis Visit Window (in study days) <sup>2, 3</sup> |
|---|---|---|---|
| Safety Assessment | | <u> </u> | · |
| Serum Chemistry | Day 1 (Baseline) | 1 | ≤1 Pre-dose |
| Hematology | Day 15 | 15 | [1, 22] |
| | Week 4 | 29 | (22, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | Use nominal visit |
| Standard 12-lead ECG | Day 1 (Baseline) | 1 | ≤1 Pre-dose |
| | Day 15 Pre-dose and | Not applicable | Use nominal visit |
| | Postdose | | |
| | Week 4 | 29 | (22, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | Use nominal visit |
| Vital Signs (excluding BMI, | Day 1 (Baseline) | 1 | ≤1 |
| Weight, Height and their Z- | Day 15 | 15 | [1, 22] |
| scores) | Week 4 | 29 | (22, 43] |
| , | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | Use nominal visit |
| Coagulation | Day 1 (Baseline) | 1 | ≤1 Pre-dose |
| C | Week 24 | 169 | [1, 183] |
| | Safety Follow-up | Not applicable | Use nominal visit |
| Efficacy Assessment and Pha | | | |
| Spirometry | Day 1 (Baseline) | 1 | ≤1 Pre-dose |
| • | Day 15 | 15 | (1, 22] |
| | Week 4 | 29 | (22, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | >183 |

| Table 12-1 Analysis Visit Windows for Safety and Efficacy Assessments | | | |
|---|---|---|---|
| Assessment | Visit <sup>1</sup> | Target Study Day | Analysis Visit Window (in study days) <sup>2, 3</sup> |
| Sweat Chloride | Day 1 (Baseline) | 1 | ≤1 Pre-dose |
| | Week 4 | 29 | (1, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 127] |
| | Week 24 | 169 | (127, 183] |
| CFQ-R | Day 1 (Baseline) | 1 | ≤1 |
| | Week 4 | 29 | (1, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | >183 |
| Weight, Height and BMI (and | Day 1 (Baseline) | 1 | ≤1 |
| the corresponding z-score) | Day 15 | 15 | (1, 22] |
| | Week 4 | 29 | (22, 43] |
| | Week 8 | 57 | (43, 71] |
| | Week 12 | 85 | (71, 99] |
| | Week 16 | 113 | (99, 141] |
| | Week 24 | 169 | (141, 183] |
| | Safety Follow-up | Not applicable | >183 |

#### Notes:

- a. If no numerical measurement is available within a visit window, the measurement will be considered missing for the visit.
- b. If there is more than 1 numerical measurement available within a visit window, use the following rules:
  - i. The measurement closest to the target day will be used; or
  - ii. If there are multiple measurements with the same distance from the target day, the latest measurement will be used.

- a. Scheduled measurement will be treated as pre-dose observation.
- b. Unscheduled measurement will be treated as post-dose observation.

#### Derived Variables:

1. Age (in years) at first dose date and nominal visit (for demographics, listing and the calculation of [percent] predicted spirometry variables):

Obtain the age at informed consent (in days) in "yy, mm" format (e.g., 24 years, 6 months) from the Vital Signs (VS) page at the Screening Visit, and add 0.5 month to convert to days.

Obtain the informed consent date.

Then age (in years) at first dose or nominal visit = [(first dose date or nominal visit date – informed consent date) in days + age at informed consent (in days)]/365.25.

<sup>&</sup>lt;sup>1</sup> Visit name for analysis purpose is used to report data in tables and figures.

<sup>&</sup>lt;sup>2</sup> The analysis visit windows will be applied using the following rules for both scheduled and unscheduled visits:

<sup>&</sup>lt;sup>3</sup> For lab, ECG and vital sign measurement collected on the date of first dose of study drug, if it cannot be determined whether the measurement is before or after the first dose:

| <b>Table 12-1</b> | Table 12-1 Analysis Visit Windows for Safety and Efficacy Assessments | | |
|---|---|---|---|
| Assessment | Visit <sup>1</sup> | Target Study Day | Analysis Visit Window (in study days) <sup>2, 3</sup> |

2. Age (in months) at nominal visit (for use in calculation of BMI and weight z-score):

Obtain the age at informed consent (in months) in "yy, mm" format (e.g., 24 years, 6 months) from Vital Signs (VS) page at the Screening Visit.

Obtain the informed consent date.

Then age (in months) at nominal visit = integer part of  $\{[(age at informed consent (in months) + 0.5 + diff(first dose date or nominal visit date, informed consent date) in months]\} + 0.5.$ 

3. Missing first dose date or last dose date

If the first dose date is missing, use Day 1 visit date to impute.

If the last dose date is missing or partial date is reported, the last dose date will be imputed based on, in descending order priority, the Early Treatment Termination (ETT) visit date, last visit date before the Safety Follow-up, or the last study drug administration date from EX SDTM domain, as appropriate. The imputation algorithm will ensure the imputed last dose date does not exceed the study participation end date.

#### 4. Sweat Chloride:

Non-missing sweat chloride concentrations from the left arm and right arm with assessment end date/time for a given arm up to 30 minutes after first dose time in treatment period will be considered for baseline.

5. Electrocardiogram:

Baseline is defined as the most recent pretreatment measurement before the first dose of study drug in the Treatment Period. If multiple ECG measurements are obtained on the same calendar day during the TE period,

- For summary purpose, the calculated average ECG will be used as the ECG value on that day (except for Day 15 visit);
- o For threshold analysis purpose, all reported ECG values will be used.
# **Appendix B: Imputation Rules for Missing Prior/Concomitant Medication Dates**

Imputation rules for missing or partial medication start/stop dates are defined below:

- 1. Missing or partial medication start date:
  - a. If only DAY is missing, use the first day of the month.
  - b. If DAY and Month are both missing, use the first day of the year.
  - c. If DAY, Month and Year are all missing, use a date before the first dose date (in practical, use Jan. 01, 2000 to impute).
- 2. Missing or partial medication stop date:
  - a. If only DAY is missing, use the last day of the month.
  - b. If DAY and Month are both missing, use the last day of the year.
  - c. If DAY, Month and year are all missing, assign 'continuing' status to stop date (in practical, use Dec. 31, 2050 to impute).

In summary, the prior, concomitant, or post categorization of a medication is described below.

Table 12-2 Prior, Concomitant, and Post Categorization of a Medication

| | | Medication Stop Date | |
|---|---|---|---|
| | < First Dose Date of<br>Study Drug | ≥ First Dose Date<br>and<br>< End Dote of TE | > End Date of TE<br>Period |
| <b>Medication Start Date</b> | | ≤ End Date of TE<br>Period | |
| < First dose date of study drug | P | PC | PCA |
| ≥ First dose date and<br>≤ End date of TE period | - | С | CA |
| > End date of TE period | - | - | A |

P: Prior; C: Concomitant; A: Post

Imputation rules for missing and/or partial dates of non-pharmacological treatment/procedure will follow the same imputation rule.

# Appendix C: Details of GLI Equations for Calculating ppFEV<sub>1</sub>

Percent predicted values will be calculated for parameters of FEV<sub>1</sub>, using the Quanjer GLI-2012 Regression Equations and Lookup Tables.

The regression equations and lookup tables required to implement the Quanjer GLI-2012 predicted values are available in:

Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Quanjer GLI-2012 Regression Equation and Lookup Tables (Version 7 April 2013). Global Lung Function Initiative. [online] Available at: http://www.ers-education.org/home/browse-all-content.aspx?idParent=138978 [Accessed Mar 26, 2018].

The instructions and tools on how to implement the Quanjer GLI-2012 equations are:

Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Implementing GLI-2012 regression equations (Version 19 July 2015). Global Lung Function Initiative. [online] Available at: http://www.ers-education.org/home/browse-all-content.aspx?idParent=138979 [Accessed Mar 26, 2018].

Sanja Stanojevic. GLI-2012 - SAS Macro (Version 2, 7 April 2013). Global Lung Function Initiative. [online] Available at: http://www.ers-education.org/home/browse-all-content.aspx?idParent=138988 [Accessed Mar 26, 2018].

Data handling rule for spirometry is as follows:

- Input age with at least 2 decimal place
- Use height at screening regardless if height is collected at other study visits for subjects whose age at informed consent is >21 years. For subjects with age <=21 years, height collected at the respective visit should be used; if the height at the respective visit is not available, the last non-missing record will be used.
- For race, map the CRF reported Black or African American to Black, all other races in CRF (except White) are mapped to 'other'; multiple checks for race in CRF are also mapped to 'other'; white is a reference race in the equations and assumes 0 values for all race coefficients in the GLI equations.

# Appendix D: Steps for Multiple Imputation

For the multiple imputation (MI) to be applied to the MMRM for the sensitivity analysis of the primary efficacy endpoint, the following steps will be followed:

### Imputation distribution

The imputation distribution for the missing absolute change from baseline in ppFEV<sub>1</sub> at visit t will be a normal distribution. All subjects in the corresponding analysis set (e.g., FAS) will be classified into one of three categories based on the following rules:

- Non-missing category: Subjects who have a ppFEV<sub>1</sub> assessment at the last timepoint of the dependent variable. Given the primary analysis method, this corresponds to the subjects who have a non-missing absolute change from baseline in ppFEV<sub>1</sub> at Week 24.
- Missing category 1: Subjects with missing absolute change from baseline in ppFEV<sub>1</sub> at the last timepoint of the dependent variable (Week 24), who discontinued treatment because of adverse events, noncompliance with study drug, death, or physician decision, or because the subject refused further dosing or required prohibited medication.
- Missing category 2: Subjects with missing absolute change from baseline in ppFEV<sub>1</sub> at the last timepoint of the dependent variable (Week 24), who completed the protocolspecified treatment or discontinued treatment for any reason not listed in Category 1.

### Imputation algorithm

We will use the following algorithm that relates the mean of the missing absolute change from baseline in ppFEV<sub>1</sub> at visit t to the missing categories defined above. The algorithm will be implemented within each treatment group as follows:

- Missing category 1: randomly draw a sample from the normal distribution  $(\mu_{25}, \sigma^2)$ , where  $\mu_{25}$  is the 25<sup>th</sup> percentile of the non-missing absolute changes from baseline in ppFEV<sub>1</sub> at visit t and  $\sigma^2$  the sample variance estimated using the non-missing absolute changes at visit t.
- Missing category 2: randomly draw a sample from the normal distribution  $(\mu, \sigma^2)$ , where  $\mu$  is the mean of the non-missing absolute changes from baseline in ppFEV<sub>1</sub> at visit t and  $\sigma^2$  is the sample variance estimated using the non-missing absolute changes at visit t.

#### **Analysis model**

The complete MI method is described below:

- Form an "imputed dataset" by imputing missing values at each visit for those subjects who have a missing value at the visit and have all subsequent values missing. The appropriate normal distribution specified in the algorithm above will be used for each such subject, based on their category.
- Repeat this process K (K=20) times to form K imputed datasets.
- Fit the same MMRM model as the one used for primary analysis to each imputed dataset to estimate the absolute change at Week 4.
- Combine the results from the analyses of K imputed datasets using the SAS procedure MIANALYZE to derive the MI estimator.

Let  $\theta$  be the true treatment difference. Denote by  $\tilde{\theta}_k$  the estimate of  $\theta$  from the  $k^{\text{th}}$  imputed dataset, and the corresponding estimate of the variance is denoted by  $V_k$ . The MI estimator of  $\theta$ ,  $\tilde{\theta}_{\text{MI}}$ , is the average of the K individual estimates.

The estimated variance of  $\tilde{\theta}_{\text{MI}}$  is a combination of the between- and within-imputation variability as follows:  $V_{\text{MI}} = W + \left(1 + \frac{1}{K}\right)B$ , where  $W = \frac{1}{K}\sum_{k=1}^{K}V_k$  is the within-imputation variability and is  $B = \frac{1}{K-1}\sum_{k=1}^{K}(\tilde{\theta}_k - \tilde{\theta}_{\text{MI}})^2$  is the between-imputation variance. The statistic  $T = \frac{\tilde{\theta}_{\text{MI}} - \theta}{\sqrt{V_{\text{MI}}}}$  has an approximate  $t_V$  distribution<sup>7</sup>, where  $V = (K-1)(1 + \frac{W}{R})^2$ .

# Appendix E: Imputation Rules for Missing AE dates

Imputation rules for missing or partial AE start date are defined below. If the imputed AE start date is before the study informed consent date, the AE start date will be imputed using the study informed consent date.

#### • If only Day of AE start date is missing:

- o If the full (or partial) AE end date is NOT before the first dose date of the Treatment Period or AE end date is missing, then
  - if AE start year and month are equal to the month and year of first dose date of the Treatment Period, then impute the AE start day as the day of first dose date of the Treatment Period:
  - else impute the AE start day as 1.
- o else impute the AE start day as 1.

Compare the imputed AE start date with TE period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

# • If Day and Month of AE start date are missing:

- o If the full (or partial) AE end date is NOT before the first dose date of the Treatment Period or AE end date is missing, then
  - if AE start year is equal to the year of first dose date of the Treatment Period, then impute the AE start month and day as the month and day of first dose date of the Treatment Period;
  - else impute the AE start month as January and day as 1.
- o else impute the AE start month as January and day as 1.

Compare the imputed AE start date with TE period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

#### • If Year of AE start date is missing:

If the year of AE start is missing or AE start date is completely missing then query site and

- If the full (or partial) AE end date is NOT before the first dose date of the Treatment Period or AE end date is missing, then impute the AE start date as the first dose date of the Treatment Period;
- o else impute the AE start date as the informed consent date.

Imputation rules for partial AE end date are defined below:

- Impute the AE end date as min (the last day of the month, end of study participation) if day is missing, or min (Dec, end of study participation) if month is missing.
  - o For the IA purpose, if the end of study date is missing, then the IA data cutoff date will be used instead in the imputation

# **Appendix F: Criteria for Threshold Analysis**

Table 12-3 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| Clinical Chemistry (LFT) | | |
| ALT | >ULN - ≤3xULN<br>>3x - ≤5xULN<br>>5x - ≤8xULN<br>>8x - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| AST | >ULN - ≤3xULN<br>>3x - ≤5xULN<br>>5x - ≤8xULN<br>>8x - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| ALT or AST | (ALT>ULN - $\leq$ 3xULN) or (AST>ULN - $\leq$ 3xULN)<br>(ALT>3x - $\leq$ 5xULN) or (AST>3x - $\leq$ 5xULN)<br>(ALT>5x - $\leq$ 8xULN) or (AST>5x - $\leq$ 8xULN)<br>(ALT>8x - $\leq$ 20xULN) or (AST>8x - $\leq$ 20xULN)<br>ALT>20xULN or AST>20xULN | FDA DILI Guidance |
| Alkaline Phosphatase | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN<br>>2.5 - ≤5.0xULN<br>>5.0 - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| Total Bilirubin | >ULN - ≤1.5xULN<br>>1.5 - ≤2xULN<br>>2 - ≤3xULN<br>>3 - ≤10xULN<br>>10xULN | FDA DILI Guidance Jul 2009. |
| Direct Bilirubin | >ULN - ≤1.5xULN<br>>1.5 - ≤2xULN<br>>2 - ≤3xULN<br>>3 - ≤10xULN<br>>10xULN | FDA DILI Guidance Jul 2009. |
| ALT and Total Bilirubin | ALT>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. |
| AST and Total Bilirubin | AST>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. |
| (ALT or AST) and Total Bilirubin | (ALT>3xULN or AST>3xULN) and TBILI>2×ULN | FDA DILI Guidance Jul 2009. |

Table 12-3 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| GGT | >ULN - ≤2.5xULN<br>>2.5 - ≤5.0xULN<br>>5.0 - ≤20.0xULN<br>>20.0xULN | CTCAE grade 1-4 |
| Clinical Chemistry (NON-LFT) | | |
| Albumin | <lln -="" g="" l<br="" ≥30="">&lt;30 - ≥20 g/L<br/>&lt;20 g/L</lln> | CTCAE grade 1-3 |
| Amylase | >1x - ≤1.5xULN<br>>1.5x - ≤2xULN<br>>2x - ≤5xULN<br>>5xULN | Criteria based upon CTCAE |
| Creatinine | >ULN - ≤1.5xULN<br>>1.5 - ≤3.0xULN<br>>3.0 - ≤6.0xULN<br>>6.0xULN | CTCAE grades 1-4 |
| Lipase | >ULN - ≤1.5xULN<br>>1.5x - ≤2xULN<br>>2x - ≤5xULN<br>>5xULN | Criteria based upon CTCAE |
| Total protein | <lln<br>&gt;ULN</lln<br> | No CTCAE |
| Creatine kinase | >ULN - ≤2.5xULN<br>>2.5 - ≤5xULN<br>>5 - ≤10xULN<br>>10xULN | CTCAE grades 1-4 |
| Hematology | | |
| Hemoglobin | Hgb decreased (anemia) <lln -="" <100="" <80="" g="" l="" l<="" td="" ≥100="" ≥80=""><td>CTCAE grade 1-3</td></lln> | CTCAE grade 1-3 |
| | Hgb increased >ULN - ≤20 g/L above ULN >20 g/L above ULN - ≤40 g/L above ULN >40 g/L above ULN | CTCAE grade 1-3 |
| Platelets | Platelet decreased<br><lln -="" 10e9="" l<br="" x="" ≥75.0="">&lt;75.0 - ≥50.0 x 10e9 /L<br/>&lt;50.0 - ≥25.0 x 10e9 /L<br/>&lt;25.0 x 10e9 /L</lln> | CTCAE grade 1-4 |
| | Platelet increased >ULN | No CTCAE available |
| Reticulocytes/Erythrocytes (%) | <lln<br>&gt;ULN</lln<br> | No CTCAE |

Table 12-3 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| Coagulation | | |
| Activated partial thromboplastin time (PTT) | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN<br>>2.5xULN | CTCAE grade 1-3 |
| Prothrombin time (PT) International Normalized Ratio (INR) | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN<br>>2.5 x ULN | CTCAE grade 1-3 |

Table 12-4 Threshold Analysis Criteria for ECGs

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| HR | Bradycardia | Per HV grade 2, 3, plus shift change |
| | <50 bpm | |
| | <45 bpm | |
| | Decrease from baseline ≥10 bpm | |
| | Decrease from baseline ≥20 bpm | |
| | <50 bpm and decrease from baseline ≥10 bpm | |
| | <50 bpm and decrease from baseline ≥20 bpm | |
| | Tachycardia | Per HV grade 1, 2, 3, plus shift change |
| | >100 bpm | |
| | >115 bpm | |
| | >130 bpm | |
| | Increase from baseline ≥10 bpm | |
| | Increase from baseline ≥20 bpm | |
| | >100 bpm and increase from baseline ≥10 bpm | |
| | >100 bpm and increase from baseline ≥20 bpm | |
| PR | ≥240 ms | |
| | ≥300 ms | |
| | ≥200 ms and increase from baseline ≥40 ms | |
| | ≥200 ms and increase from baseline ≥100 ms | |
| QRS | >110 ms | |
| | >160 ms | |
| | Increase from baseline ≥20 ms | |
| | Increase from baseline ≥40 ms | |
| QTc | >450 to <500ms (Male) or >470 to <500ms (Fema | |
| | ≥500 ms | correction formula. |
| | Increase from baseline | |
| | Increase from baseline >10 ms | |
| | Increase from baseline >20 ms | |
| | Increase from baseline >40 ms | |
| | Increase from baseline >60 ms | |

Table 12-5 Threshold Analysis Criteria for Vital Signs

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| Pulse Rate | Same as above in ECG category | |
| SBP increased | >140 mmHg<br>>160 mmHg<br>>10 mmHg increase from baseline<br>>20 mmHg increase from baseline | 809/770 analyses |
| | >140 mmHg & >10 mmHg increase from baseline<br>>140 mmHg & >20 mmHg increase from baseline<br>>160 mmHg & >10 mmHg increase from baseline<br>>160 mmHg & >20 mmHg increase from baseline | |
| SBP decrease | <90 mmHg<br><80 mmHg<br>>10 mmHg decrease from baseline<br>>20 mmHg decrease from baseline | Per HV grade 1, 3, plus shift change |
| | <90 mmHg and >10 mmHg decrease from baseline<br><90 mmHg and >20 mmHg decrease from baseline<br><80 mmHg and >10 mmHg decrease from baseline<br><80 mmHg and >20 mmHg decrease from baseline | |
| DBP increased | >90 mmHg<br>>100 mmHg<br>>5 mmHg increase from baseline<br>>10 mmHg increase from baseline | |
| | >90 mmHg and >5 mmHg increase from baseline<br>>90 mmHg and >10 mmHg increase from baseline<br>>100 mmHg and >5 mmHg increase from baseline<br>>100 mmHg and >10 mmHg increase from baseline | |
| DBP decreased | <60 mmHg<br><45 mmHg<br>>5 mmHg decrease from baseline<br>>10 mmHg decrease from baseline | |
| | <60 mmHg and >5 mmHg decrease from baseline<br><60 mmHg and >10 mmHg decrease from baseline<br><45 mmHg and >5 mmHg decrease from baseline<br><45 mmHg and >10 mmHg decrease from baseline | |
| Weight | Weight gain ≥5 % increase from baseline ≥10 % increase from baseline ≥ 20% increase from baseline | CTCAE grade 1-3 |
| | Weight loss ≥5 % decrease from baseline ≥10 % decrease from baseline ≥ 20% decrease from baseline | CTCAE grade 1-3 |

Table 12-6 Threshold Analysis Criteria for Laboratory Tests (for labeling purpose)

| Parameter | Threshold Analysis | Comments |
|------------------------|--------------------|----------------------|
| Clinical Chemistry (LF | TT) | |
| ALT or AST | >3xULN | For labeling purpose |
| | >5xULN | |
| | >8xULN | |

# **Appendix G: Adverse Events of Special Interest**

| Table 12-7 MedDRA Preferred Terms for Event of Special Interest | |
|---|---|
| Adverse event of special interest | MedDRA preferred terms |
| Elevated transaminase | Alanine aminotransferase abnormal, Alanine aminotransferase increased, Aspartate aminotransferase abnormal, Aspartate aminotransferase increased, Transaminases abnormal, Transaminases increased, Liver function test abnormal, Liver function test increased, Hypertransaminasaemia, Hepatic enzyme abnormal, Hepatic enzyme increased |
| Rash | Rash, Rash erythematous, Rash macular, Rash maculo-papular, Rash maculovesicular, Rash vesicular, Rash pruritic, Rash follicular, Rash pustular, Rash generalized, Nodular rash, Drug eruption, Fixed eruption, Generalised erythema, Urticaria, Urticaria popular, Urticaria vesiculosa, Rash morbilliform, Rash popular, Rash papulosquamous, Rash rubelliform, Rash scarlatiniform, Drug hypersensitivity, Type IV hypersensitivity reaction, Dermatitis, Dermatitis atopic, Epidermolysis, Skin toxicity, Dermatitis allergic, Dermatitis exfoliative, Dermatitis exfoliative generalized, Erythema multiforme, Exfoliative rash, Mucocutaneous rash, Acute generalised exanthematous pustulosis, Cutaneous vasculitis, Urticarial vasculitis, Dermatitis bullous, Drug reaction with eosinophilia and systemic symptoms, Epidermal necrosis, Oculomucocutaneous syndrome, Skin exfoliation, Skin necrosis, Stevens-Johnson syndrome, Toxic epidermal necrolysis, Toxic skin eruption, Perioral dermatitis, Vasculitic rash |

Note: the preferred terms listed in the table is based on the MedDRA version applicable at the time of finalization of the SAP. If the MedDRA version is upgraded at the time of the analysis, the corresponding preferred terms based on the upgraded version will be used in the analysis of adverse events of special interest.

#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Addendum to Statistical Analysis Plan (Methods)

Protocol Number VX17-445-102 Version 3.0 (Final and Interim Analysis)

A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the *F508del* Mutation and a Minimal Function Mutation (F/MF)

**Authors of SAP:** 

Version: 1.0

Version Date of Addendum: 17 December 2018 Version Date of SAP: 25 September 2018

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, Massachusetts 02210-1862


This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Addendum 2 to Statistical Analysis Plan (Methods)

Protocol Number VX17-445-102 Version 3.0 (Final Analysis)

A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the *F508del* Mutation and a Minimal Function Mutation (F/MF)

**Authors of Addendum 2:** 



Version of Addendum 2: 1.0 Version Date of Addendum 2: 21MAR2019

**Original Version Date of SAP: 25SEP2018** 

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, Massachusetts 02210-1862


This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# 2 TABLE OF CONTENTS

| 1 | Tit | le Page |
|---|---|---|
| | Table of Contents | |
| | Modifications | |
| | | Modifications to the Approved Clinical Study Protocol |
| | | Modifications to the Approved Statistical Analysis Plan |
| | | Modifications to the Approved Addendum |
| | Introduction | |
| | 5 Statistical Analysis | |
| | | General Considerations |
| | 5.2 | Efficacy Analysis |
| | 5.2.1 Analysis of Endpoints Based on the Number of Clinical Events | |

# 3 MODIFICATIONS

# 3.1 Modifications to the Approved Clinical Study Protocol

Not Applicable.

# 3.2 Modifications to the Approved Statistical Analysis Plan

Not Applicable.

# 3.3 Modifications to the Approved Addendum

This is the 1<sup>st</sup> version of Addendum 2 to the statistical analysis plan for the final analysis. There is no change to the preceding Addendum 1 which was approved on 17DEC2018.

Protocol Number: VX17-445-102

#### 4 INTRODUCTION

This Addendum 2 to the statistical analysis plan (SAP) for the final analysis is based on the approved SAP (Version 1.0, approval date: 25SEP2018; Version 1.1 EUR approval date: 10DEC2018), as well as the preceding Addendum 1 (Version 1.0, approval date: 17DEC2018).

Addendum 2 documents additional statistical analyses for selected efficacy variables for the final analysis. This addendum will be finalized and approved prior to the final database lock. Any revisions to the approved addendum will be documented and approved as a new version of the addendum.

The Vertex Biometrics Department will perform the additional analyses specified in this Addendum 2 for the final analysis; SAS (Version 9.4 or higher) will be used to generate all statistical outputs (tables, figures, listings, and datasets).

#### 5 STATISTICAL ANALYSIS

This section discusses the additional analyses planned for the final analysis.

#### 5.1 General Considerations

No change to the general considerations specified in the SAP.

# 5.2 Efficacy Analysis

#### 5.2.1 Analysis of Endpoints Based on the Number of Clinical Events

Number of Pulmonary Exacerbation (PEx) through Week 24: The analysis pre-specified in the protocol based on the negative binomial regression model will be performed first. If the negative binomial regression does not converge, the analysis will be performed using the Poisson regression with the same covariates and offset.

Note: If the number of events is less than 5 in either treatment group, neither the negative binomial regression nor the Poisson regression will be performed and analysis of event counts will be based on a Fisher's Exact test.

Analysis of the number of PEx requiring hospitalization and/or IV antibiotics therapy, the number of planned hospitalizations for CF, and the number of unplanned hospitalizations for reasons other than antibiotic therapy for sinopulmonary signs/symptoms will be performed in the same manner.